CLINICAL TRIAL: NCT00941187
Title: Evolution of Pulmonary Capillary Blood Volume (Vc) in Patients After a First Episode of Pulmonary Embolism.
Brief Title: Evolution of Pulmonary Capillary Blood Volume
Acronym: VcEP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0808076; 2008-A01122-53 (Other: AFSSAPS)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary embolism; pulmonary capillary blood volume; double diffusion NO/CO method
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients after a first episode of pulmonary embolism
  Interventions: Other: diffusion NO/CO method

INTERVENTIONS:
Other: diffusion NO/CO method — pulmonary capillary blood volume (Vc), measured by the double diffusion NO/CO method: this method is to inhale during a deep inspiration with a mixture of helium (8-10%), CO (2000 ppm) and NO (20-40 ppm), the O2 (21%)

SUMMARY:
The purpose of this monocentric, preliminary study is to assess the evolution of pulmonary capillary blood volume (Vc), measured by the double diffusion nitric oxide/carbon monoxide (NO/CO) method (Guenard et al.; Respir Physiol 1987), from the starting of the anticoagulant therapy to 6 months after, and to search correlations with the evolution of clinical (dyspnea and results of the 6 minutes walking test), biological (BNP; Troponin), echocardiographic (right ventricular dysfunction, pulmonary arterial pressure) and ventilation/perfusion lung scan data.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a first episode of symptomatic pulmonary embolism, treated with anticoagulant
* Age from 18 to 75 years-old

Exclusion Criteria:

* Confirmed pulmonary embolism in the past
* Massive pulmonary embolism, thrombolytic treatment
* Confirmed left heart systolic dysfunction
* Confirmed asthma, chronic obstructive pulmonary disease or pulmonary fibrosis
* Expected life below 6 months
* Pleural effusion with indication of evacuation
* Bronchopulmonary cancer
* Pulmonary surgery with resection of two lobes minimum
* Predictable incapacity to complete the 6 minutes walking test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a first episode of symptomatic pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
difference of pulmonary capillary blood volume (Vc) from J0 to 6 months | from the starting of the anticoagulant therapy to 6 months after

SECONDARY OUTCOMES:
correlations with the evolution of clinical (dyspnea and results of the 6 minutes walking test), biological (BNP; Troponin), echocardiographic (right ventricular dysfunction, pulmonary arterial pressure) and ventilation/perfusion lung scan data | from the starting of the anticoagulant therapy to 6 months after

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BERTOLETTI, MD, Principal Investigator — CHU de Saint-Etienne
Locations (2):
- France (2):
  - Departement of pneumology, CHU Saint-Etienne, Saint-Etienne
  - Department of Medicine and Therapeutic, CHU Saint-Etienne, Saint-Etienne